CLINICAL TRIAL: NCT04934826
Title: Comparison of the Absorption of Hydrolyzed or Intact Proteins in Morbid Obese
Brief Title: Comparison of the Absorption of Hydrolyzed or Intact Proteins in Morbid Obese Patients After the Roux Y Gastric Bypass
Acronym: RyDIGEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D20180131; 2019-A01448-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-02-24; First posted 2021-06-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrolized proteins (Experimental): Group receiving hydrolyzed proteins in the postprandial metabolic test
  Interventions: Dietary Supplement: Hydrolyzed Proteins
- Intact proteins (Active Comparator): Group receiving intact proteins in the postprandial metabolic test
  Interventions: Dietary Supplement: Intact proteins

INTERVENTIONS:
Dietary Supplement: Hydrolyzed Proteins — Patients in experimental arm will receive a test meal based on marked hydrolyzed proteins
  Arms: Hydrolized proteins
Dietary Supplement: Intact proteins — Patients in active comparator arm will receive a meal based on intact marked proteins.
  Arms: Intact proteins

SUMMARY:
The gastric bypass can reduce the bioavailability of food proteins. The bioavailability of hydrolyzed proteins may be higher than intact proteins. Thus, the use of hydrolyzed proteins could compensate for the decrease in protein bioavailability observed after gastric By-pass in morbidly obese patients.

The effectiveness of a hydrolyzed protein intake may be higher than that of an intact protein intake to improve the status of a By-pass.

The hypothesis would be that the use of hydrolyzed proteins would compensate for the decrease in bioavailability of food proteins caused by gastric By-pass.

DETAILED DESCRIPTION:
Surgery is beneficial in terms of weight loss, correction of comorbidities and life expectancy but adverse effects can occur among which various nutritional deficiencies. Thus, in some cases, more or less marked protein undernutrition may be observed.

To overcome this protein undernutrition, protein supplements can be proposed. However, their effectiveness has not been satisfactorily assessed in this situation to date. Indeed, the protein malabsorption potentially induced by the By-pass limits its impact. The value of protein supplementation must also be considered in terms of overall efficacy, taking into account a possible decrease in spontaneous intake related to supplementation.

For the bioavailability studies, milk proteins will be presented in two different forms of the same origin: intact or hydrolyzed proteins. The proteins of the test meal are marked with 15N nitrogen.

For the three months daily supplementation period, the supplements will be intact proteins not marked with 15N nitrogen, provided to patients in the form of individual sachets. The purpose of this supplementation is to help the patient achieve the protein recommendations, which is 60 g/d.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with BMI > 40 kg/m2 or BMI > 35 kg/m2 associated with at least one comorbidity(s): hypertension, diabetes, cardiovascular disease, hyperlipidemia, sleep apnea, arthritis,hepatic steatosis.
2. Candidates for RY gastric By-pass bariatric surgery,
3. Over 18 and under 60 years of age
4. For women of childbearing age: effective contraception implemented for at least 3 months.
5. Failure of other medical cares (medical, nutritional, dietetic and psychotherapeutic treatment) well conducted for 6 to 12 months.
6. Patient affiliated to a social security system (excluding AME) or entitled to benefits.
7. Patient who agreed to participate by signing the informed consent of the study

Exclusion Criteria:

1. Pregnancy or breastfeeding in progress
2. Severe psychiatric disorder or other illness that may disrupt the study follow-up or to invalidate the proper understanding of the protocol information and the informed consent
3. Patient's foreseeable inability to participate in a clinical trial
4. Severe and unstable eating disorders
5. Patients with a contraindication to amino acid infusion
6. Dependence on alcohol or psychoactive substances such as drugs
7. Metabolic disease requiring a a low protein diet
8. Known allergy to milk proteins
9. Patient under guardianship or curatorship
10. Patient under the justice protection
11. Participation in another interventional research

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Compare the evolution of the bioavailability of hydrolyzed milk proteins to the intact milk proteins in obese patients who have received a By-pass, using the Nitrogen-15 (15N) labelled test meal method | 6 months after By-pass
  The evolution of bioavailability will be evaluated by the delta of post-prandial bioavailability of food proteins (hydrolysed vs intact) before and 6 months after By-pass.

SECONDARY OUTCOMES:
Evaluate the effect of daily milk protein supplementation administered for 3 months after a post-surgery recovery period of 3 months on protein status in obese patients who had a By-pass. | 6 months after By-pass
  The effect of an intact milk protein supplementation, administered between 3 months and 6 months after the By-pass, will be evaluated by the variation of albuminemia measured by DEXA and by impedancemetry before 3 months and 6 months after By-pass.
  he effect of an intact milk protein supplementation, administered between 3 months and 6 months after the By-pass, will be evaluated by the variation of pre-albuminemia measured by DEXA and by impedancemetry before 3 months and 6 months after By-pass.
  he effect of an intact milk protein supplementation, administered between 3 months and 6 months after the By-pass, will be evaluated by the variation of lean mass measured by DEXA and by impedancemetry before 3 months and 6 months after By-pass.
Evaluate the compliance with supplementation of an intact milk protein administered for 3 months after a post-surgery recovery period of 3 months, in obese patients who had a By-pass, as well as its contribution to daily protein intake. | 6 months after By-pass
  The compliance of an intact milk protein supplementation, administered between 3 months and 6 months after the By-pass, will be evaluated by the variation in food intake and protein intake, determined in a food survey
Evaluate the compliance with supplementation of an intact milk protein administered for 3 months, after a post-surgery recovery period of 3 months, on spontaneous food consumption in obese patients who had a By-pass. | 6 months after By-pass
  The compliance of an intact milk protein supplementation, administered between 3 months and 6 months after the By-pass, will be evaluated by the variation in food intake and protein intake.
Evaluate the effect of an intact milk protein supplementation administered for 3 months after a post-surgery recovery period of 3 months, on the quality of life in obese patients who have undergone a By-pass surgery. | 6 months after By-pass
  The effect of administered an intact protein supplementation between 3 months and 6 months after the By-pass on quality of life will be assessed using the Obesity Weight Loss Quality of Life (OWLQOL).
Evaluate post-prandial splanchnic sequestration of dietary amino acids | 6 months after By-pass
  The transfer of 15N nitrogen is evaluated after determination of the enrichment by isotope ratio mass spectrometry (IRMS), the main endpoint is the rate of transfer of 15N nitrogen into the metabolic pools: plasma proteins, plasma urea and urine. In addition, the 15N and 13C isotopic ratios will be determined in the individual blood amino acids by mass spectrometry coupled with gas and combustion chromatography (GC-c-IRMS), in order to determine the digestive bioavailability of the amino acids of the proteins of the test meal.
Evaluate the effect of an intact milk protein supplementation administered for 3 months after a post-surgery recovery period of 3 months, on the quality of life in | 6 month
  he effect of administered an intact protein supplementation between 3 months and 6 months after the By-pass on quality of life will be assessed using the Weight-Related Symptom Measure (WRSM) questionnary.

CONTACTS AND LOCATIONS:
Overall Officials: Gheorghe AIRINEI, Doctor, Principal Investigator — Assistance Publique - Hôpitaux Paris
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: The final report of the research will be drawn up and signed by the sponsor and the investigator.
  A summary of the report drawn up according to the reference plan of the competent authority will be sent to the competent authority within one year so it will be sent on february, 2025, after the end of the research, corresponding to the end of the participation of the last person who is willing.
Access Criteria: The access criteria IPD and any additional supporting information will be shared in the final report or publication. The analysis will be carried out on a modified intention-to-treat basis: all included patients, randomized and whose evaluation at 6 months after surgery will be available, will participate in the analysis in the group assigned by the random draw. This analysis avoids taking into account the patients who will be lost to follow-up before the evaluation at 6 months after the intervention. A per-protocol analysis will also be carried out. Changes in study weight, body composition, blood markers and food intake will be compared between groups using a mixed repeated measures model, with group as a fixed effect and time as the intra-repeat factor. topic. The group's effect on quality of life scores will be analyzed using a Wilcoxon test.

REFERENCES:
- [Background] Airinei G, Gaudichon C, Bos C, Bon C, Kapel N, Bejou B, Raynaud JJ, Luengo C, Aparicio T, Levy P, Tome D, Benamouzig R. Postprandial protein metabolism but not a fecal test reveals protein malabsorption in patients with pancreatic exocrine insufficiency. Clin Nutr. 2011 Dec;30(6):831-7. doi: 10.1016/j.clnu.2011.06.006. Epub 2011 Jul 8. PMID 21741734
- [Background] Aron-Wisnewsky J, Verger EO, Bounaix C, Dao MC, Oppert JM, Bouillot JL, Chevallier JM, Clement K. Nutritional and Protein Deficiencies in the Short Term following Both Gastric Bypass and Gastric Banding. PLoS One. 2016 Feb 18;11(2):e0149588. doi: 10.1371/journal.pone.0149588. eCollection 2016. PMID 26891123
- [Background] Bos C, Airinei G, Mariotti F, Benamouzig R, Berot S, Evrard J, Fenart E, Tome D, Gaudichon C. The poor digestibility of rapeseed protein is balanced by its very high metabolic utilization in humans. J Nutr. 2007 Mar;137(3):594-600. doi: 10.1093/jn/137.3.594. PMID 17311946
- [Background] Bos C, Juillet B, Fouillet H, Turlan L, Dare S, Luengo C, N'tounda R, Benamouzig R, Gausseres N, Tome D, Gaudichon C. Postprandial metabolic utilization of wheat protein in humans. Am J Clin Nutr. 2005 Jan;81(1):87-94. doi: 10.1093/ajcn/81.1.87. PMID 15640465
- [Background] Oberli M, Marsset-Baglieri A, Airinei G, Sante-Lhoutellier V, Khodorova N, Remond D, Foucault-Simonin A, Piedcoq J, Tome D, Fromentin G, Benamouzig R, Gaudichon C. High True Ileal Digestibility but Not Postprandial Utilization of Nitrogen from Bovine Meat Protein in Humans Is Moderately Decreased by High-Temperature, Long-Duration Cooking. J Nutr. 2015 Oct;145(10):2221-8. doi: 10.3945/jn.115.216838. Epub 2015 Aug 19. PMID 26290008
- [Background] Lacroix M, Bos C, Leonil J, Airinei G, Luengo C, Dare S, Benamouzig R, Fouillet H, Fauquant J, Tome D, Gaudichon C. Compared with casein or total milk protein, digestion of milk soluble proteins is too rapid to sustain the anabolic postprandial amino acid requirement. Am J Clin Nutr. 2006 Nov;84(5):1070-9. doi: 10.1093/ajcn/84.5.1070. PMID 17093159
- [Background] Boutrou R, Gaudichon C, Dupont D, Jardin J, Airinei G, Marsset-Baglieri A, Benamouzig R, Tome D, Leonil J. Sequential release of milk protein-derived bioactive peptides in the jejunum in healthy humans. Am J Clin Nutr. 2013 Jun;97(6):1314-23. doi: 10.3945/ajcn.112.055202. Epub 2013 Apr 10. PMID 23576048
- See also: Guide written by French Food Safety Agency about "Protein intake: consumption, quality, needs and recommendations" — https://www.anses.fr/fr/system/files/NUT-Ra-Proteines.pdf